CLINICAL TRIAL: NCT03974321
Title: Association Between Intraoperative Hypotension and Perioperative Myocardial Injury: a Nested Case Control Study
Brief Title: Intraoperative Hypotension and Perioperative Myocardial Injury
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Max Bell, MD, PhD, Associate Professor, Senior Lecturer, Karolinska Institutet
Other Study IDs: 20180713
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Myocardial Infarction Postoperative; Myocardial Injury; Intraoperative Complications; Intraoperative Hypotension; Perioperative Complication
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute myocardial infarction (MI) is a significant complication following non-cardiac surgery. We sought to evaluate incidence of perioperative MI, its preoperative - and intraoperative - risk factors and outcomes after this complication.

DETAILED DESCRIPTION:
Background:

In Sweden, over 800 000 patents undergo surgery each year. Worldwide, the number of surgical procedures yearly is over 310 million. Surgical care is en essential part of the advancement in treating disease, associated with increased lift expectancy a d improved quality of life. However as surgical volume continues to grow, the number of patients who suffer postoperative complications will also increase.

Hemodynamic instability in the perioperative period is frequent and there has been a cumulative interest in this area and the relation to organ failure over the recent years. There are several studies showing results of associations between intraoperative hypotensive events and perioperative cardiac, kidney and cerebral injury, as well as increased mortality in high-risk surgical patients.

More specifically the project aims to answer how intraoperative events, with a special focus on hypotension, are related to perioperative myocardial and kidney injury.

We hypothesize that patients, with preoperative risk factors, undergoing major non-cardiac surgery are at increased risk of developing perioperative organ damage in the presence of intraoperative hypotension or other events such as tachycardia, hypoxia and extensive blood loss.

ELIGIBILITY:
Cases

Inclusion Criteria:

* Adults (≥18 years), male and female.
* Undergoing elective or non-elective in-patients non-cardiac surgery at 3 University Hospitals in Sweden: Karolinska University hospital, Skåne University hospital and Norrland University hospital.
* Surgeries performed between 2007 and 2014.
* Acute myocardial infarction criteria fulfilled within 30 days after surgery.

Exclusion Criteria:

* Cardiac surgery
* Obstetric surgery

Controls:

Matched (on age, preoperative risk factors, surgical year- site and procedure) surgical patients without myocardial infarction within 30 days after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing non-cardiac surgery between 2007 and 2014 at 3 Swedish University hospitals; Karolinska University hospital, Skåne University Hospital and Norrland University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Acute Myocardial Infarction | Within 30 days after the index surgery
  Acute MI, detected in the postoperative phase in the electronic medical records or in the Swedeheart Registry

SECONDARY OUTCOMES:
Mortality | Witis 30 days after the index surgery and at later predefined time points: 60, 90 180 and 365 days after the index surgery.
  Death, detected in the postoperative phase in the Swedish Cause of Death Register.

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, MD, PhD, Principal Investigator — Karolinska University Hospital, Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden